CLINICAL TRIAL: NCT02461745
Title: A Phase IV, Multisite Study of the Treatment of Chronic Hepatitis C Virus Infection Genotype 1 in a Real World Large Health Maintenance Organization: An Evaluation of Real World Sustained Virological Response and Patient Reported Outcomes
Brief Title: Real World Study: Genotype 1 Chronic Hepatitis C Virus Treatment and Evaluation of Real World SVR and PRO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KPSC IRB 10568
Record Dates: First submitted 2015-05-31; First posted 2015-06-03 (Estimated); Results first posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Hepatitis C, Chronic
Keywords: VIEKIRA PAK
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — ombitasvir; dasabuvir; Ribavirin; Viekira Pak

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Genotype 1a (Active Comparator): Study participants with chronic Hepatitis C Genotype 1A receiving VIEKIRA PAK (two 12.5/75/50 mg ombitasvir, paritaprevir, ritonavir tablets, and two 250 mg dasabuvir tablets) and RBV (ribavirin tablets) for 12 weeks.
  Interventions: Drug: ombitasvir, paritaprevir/r, dasabuvir + ribavirin
- Genotype 1b (Active Comparator): Study participants with chronic Hepatitis C Genotype 1B receiving VIEKIRA PAK (two 12.5/75/50 mg ombitasvir, paritaprevir, ritonavir tablets, and two 250 mg dasabuvir tablets) for 12 weeks.
  Interventions: Drug: ombitasvir, paritaprevir/r, dasabuvir

INTERVENTIONS:
Drug: ombitasvir, paritaprevir/r, dasabuvir + ribavirin — VIEKIRA PAK (two 12.5/75/50 mg ombitasvir, paritaprevir, ritonavir tablets, and two 250 mg dasabuvir tablets) + RBV (ribavirin tablets) for 12 weeks
  Other Names: VIEKIRA PAK + RBV
  Arms: Genotype 1a
Drug: ombitasvir, paritaprevir/r, dasabuvir — VIEKIRA PAK (two 12.5/75/50 mg ombitasvir, paritaprevir, ritonavir tablets, and two 250 mg dasabuvir tablets)
  Other Names: VIEKIRA PAK
  Arms: Genotype 1b

SUMMARY:
This is a Phase IV, open-label, multi-center study to evaluate the real world sustained virological response rate, subject adherence, and subject reported outcomes during and after treatment of non-cirrhotic genotype 1 chronic hepatitis C subjects aged 18 years and older, with VIEKIRA PAK (ombitasvir, paritaprevir/r, dasabuvir), with or without RBV (ribavirin).

DETAILED DESCRIPTION:
This is a Phase IV, open-label, multi-center study to evaluate the real world sustained virological response rate, subject adherence, and subject reported outcomes during and after treatment of non-cirrhotic genotype 1 chronic hepatitis C subjects aged 18 years and older, with the AbbVie 3 direct-acting antiviral (3-DAA) regimen of VIEKIRA PAK (ombitasvir, paritaprevir/r, dasabuvir), with or without RBV (ribavirin).

Subjects may be treatment-naïve or treatment experienced with pegylated-interferon based regimens excluding regimens with direct-acting antiviral agents. The study will be conducted at multiple Kaiser Permanente Southern California Medical Centers.

The primary objective of this open label study is to evaluate the rate of sustained virological response rate 12 weeks after completion of treatment (SVR12) with VIEKIRA PAK, with or without ribavirin in a large real world setting.

ELIGIBILITY:
Key Inclusion Criteria

* Male or female at least 18 years of age at time of screening.
* Subject, if female must not use estrogen-containing hormonal contraception including oral, injectable, implantable, patch and ring varieties during study drug treatment
* Subject, if male, who is not surgically sterile and is sexually active with female partner of childbearing potential must agree to practice 2 effective contraceptive methods for study duration
* Subject must have at least one of the following indicators of chronic hepatitis C virus infection prior to study enrollment: Positive anti-HCV antibody or HCV RNA > 10,000 IU/mL at least 6 months before screening, and positive for HCV RNA at the time of screening, or HCV RNA > 10,000 IU/mL at screening and liver biopsy consistent with chronic HCV infection
* Subject has a screening laboratory result indicating HCV genotype 1-infection

Key Exclusion Criteria

* Subject, if female is pregnant or is breastfeeding, of if male, with female partner who is currently pregnant
* Subject has positive test result for hepatitis B surface antigen or confirmed positive anti-HIV antibody test
* Subject received study contraindicated medications prior to study drug administration
* Use of known strong inducers of cytochrome P450 3A (CYP3A) or strong inducers of cytochrome P450 2C8 (CYP2C8) or strong inhibitors of CYP2C8 within 2 weeks of the respective medication/supplement prior to initial dose of study drug.
* Clinically significant abnormalities or co-morbidities, other than HCV infection that in opinion of the investigator makes subject unsuitable for this study or drug regimen
* Current enrollment in another interventional clinical study or prior or current use of any investigational or commercially available anti-HCV agents other than interferon or ribavirin including previous exposure to ABT450 (paritaprevir) , ABT-267 (ombitasvir) or ABT-333 (dasabuvir) or receipt of any investigational product within 6 weeks prior to study drug administration
* Prior treatment of chronic HCV infection with a direct acting antiviral agent(s): telaprevir, boceprevir, sofosbuvir, simeprevir, or other direct acting antiviral
* History of solid organ transplant
* Evidence of cirrhosis
* History of liver decompensation: ascites noted on a physical exam, imaging or other test; variceal bleeding; hepatic encephalopathy
* Confirmed presence of hepatocellular carcinoma indicated on computed tomography, magnetic resonance, or other imaging techniques within 3 months prior to screening
* HCV genotype performed during screening indicates infection with any genotype other than genotype 1
* Recent history of drug or alcohol abuse that could, in the opinion of the investigator, affect adherence to the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-06; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Nyberg, MD, Principal Investigator — Kaiser Permanente
Locations (4):
- United States (4):
  - Kaiser Permanente Medical Center, Irvine, California
  - Kaiser Permanente Medical Center, Los Angeles, California
  - Kaiser Permanente Medical Center, San Diego, California
  - Kaiser Permanente Medical Center, San Marcos, California

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period started in June 2015 until October 2016 at four (4) different Kaiser Permanente Southern California medical clinics.
Pre-assignment Details: 228 study participants screened for the study had 28 days from signing the study consent form to their first dose of study drug to confirm their eligibility to continue with the study. The screening period was also used as a wash-out period for concomitant medications that may interact with the study drug.
Groups:
- Genotype 1a: Study participants with chronic Hepatitis C Genotype 1a receiving VIEKIRA PAK and Ribavirin for 12 weeks.
- Genotype 1b: Study participants with chronic Hepatitis C Genotype 1b receiving VIEKIRA PAK for 12 weeks.
Period: Overall Study
Arm/Group | Genotype 1a | Genotype 1b
Started | 130 | 70
Completed | 116 | 66
Not Completed | 14 | 4
Not completed — Lack of Efficacy | 9 | 1
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrawal by Subject | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Genotype 1a | Genotype 1b | Total
Number analyzed (Participants) | 130 | 70 | 200
Age, Continuous [Mean (Full Range); unit: years] | 56.64 [20 to 75] | 60.87 [23 to 79] | 58.12 [20 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 31 | 80
  Male | 81 | 39 | 120
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 6 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 5 | 7
  White | 121 | 56 | 177
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 130 | 70 | 200
Baseline HCV RNA [Count of Participants; unit: Participants]
  <800,000 IU/mL | 27 | 17 | 44
  Between 800,000 - 6 million | 74 | 43 | 117
  >6 million | 29 | 10 | 39
Treatment-experience [Count of Participants; unit: Participants]
  Experienced | 22 | 9 | 31
  Naive | 108 | 61 | 169

OUTCOME MEASURES:

1. Primary Outcome: Sustained Virological Response (SVR) at Week 12
Description: Percentage of study participants achieving sustained virological response (SVR) at Week 12 per protocol among study participants who completed 12-week course of treatment.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Genotype 1a | Genotype 1b
Number analyzed (Participants) | 123 | 67
Participants | 116 | 66

2. Secondary Outcome: Sustained Virological Response (SVR) at Week 4
Description: Percentage of study participants achieving sustained virological response (SVR) at Week 4 per protocol among subjects who completed 12-week course of treatment in the study.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Genotype 1a | Genotype 1b
Number analyzed (Participants) | 122 | 66
Participants | 116 | 65

ADVERSE EVENTS:
Time Frame: Adverse events are collected from enrolled study participants during the treatment period (12 weeks) through an additional 12 weeks post treatment. For enrolled study participants that discontinued from the study, adverse events are collected during the treatment period until their last completed study visit.
Description: Adverse events reported in the table below are those that are considered possibly or definitely related to the VIEKIRA PAK (ombitasvir, paritaprevir/r, dasabuvir) and/or RBV (ribavirin tablets). Although adverse events data was collected from all subjects who receive at least one dose of the study drug regardless of their relationship to either VIEKIRA PARK and/or RBV, the analysis of the safety data was focused on those that are treatment-related, which is provided below.
Arm/Group | Genotype 1a | Genotype 1b
All-Cause Mortality (participants affected / at risk) | 0/130 | 0/70
Serious Adverse Events (participants affected / at risk) | 4/130 | 3/70
Other Adverse Events (participants affected / at risk) | 102/130 | 30/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Genotype 1a (N=130) | Genotype 1b (N=70)
Acute Congestive Heart Failure (Cardiac disorders) | 1 (1) | 0 (0)
Acute Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acute Psychosis (Psychiatric disorders) | 1 (1) | 0 (0)
Cellulitis/ Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Guillain Barre Syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Small Cell Carcinoma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urothelial Carcinoma (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Genotype 1a (N=130) | Genotype 1b (N=70)
Fatigue (Musculoskeletal and connective tissue disorders) | 35 (35) | 10 (10)
Nausea (Gastrointestinal disorders) | 20 (20) | 4 (4)
Headache (Nervous system disorders) | 16 (16) | 5 (5)
Insomnia (Nervous system disorders) | 13 (13) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 5 (5) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (7) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 6 (6) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-01): https://cdn.clinicaltrials.gov/large-docs/45/NCT02461745/Prot_SAP_000.pdf